CLINICAL TRIAL: NCT03764371
Title: A Prospective, Single-center, Phase II Clinical Study of the Effects of Different Genetic Mutations on Prognosis in Multiple Primary Nodular Lung Adenocarcinoma Patients
Brief Title: Effects of Different Genetic Mutations on Prognosis in sMPLC Adenocarcinoma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: K2018108
Record Dates: First submitted 2018-11-28; First posted 2018-12-05 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-08

CONDITIONS: Gene Mutation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We use application of NGS technology to test lung cancer related genes in patients' tumor tissues and blood, patients with lung cancer drive genes were followed up to explore whether different drive genes had an impact on patients' disease progression.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sMPLC: Lung cancer related genes in tumor tissues and patients with at least 2 tumors that were confirmed as invasive adenocarcinoma by pathology after sMPLC resection (residual non-resectable or non-qualitative pulmonary nodules).
  Interventions: Diagnostic Test: KAPA Hyper Prep Kit + Agilent SureSelectQXT

INTERVENTIONS:
Diagnostic Test: KAPA Hyper Prep Kit + Agilent SureSelectQXT — We initiated this prospective clinical study to detect lung cancer related genes in tumor tissues and patients with at least 2 tumors that were confirmed as invasive adenocarcinoma by pathology after sMPLC resection (residual non-resectable or non-qualitative pulmonary nodules). At the same time, application of KAPA Hyper Prep Kit + Agilent SureSelectQXT technology to test lung cancer related genes in patients' tumor tissues and blood, patients with lung cancer drive genes were followed up to explore whether different drive genes had an impact on patients' disease progression. In order to investigate the type of gene that causes disease recurrence in patients, tissue or blood test was performed again when disease recurrence occur.
  Other Names: NGS technology

SUMMARY:
In 2007 and 2013, the American College of Chest Physicians (ACCP) guidelines applied the diagnostic criteria of sMPLC （synchronous multiple primary lung cancers）, and the diagnostic criteria of Martini and Melamed were extended and developed, Summarized as: (1) different histological types, different genetic characteristics, or different origin of carcinoma in situ; (2) the histological type is the same, the tumor is located in different lung or different lung lobes, the common lymphatic drainage site of lung cancer is not cancerous, and there is no extrapulmonary metastasis at the time of diagnosis.

Postoperative staging of each tumor was carried out in sMPLC patients, if all of them were stage I lung adenocarcinoma, whether adjuvant therapy could fully refer to the treatment principle of stage I NSCLC was considered, whether the benefit of subsequent application of adjuvant chemotherapy was still unclear, and whether adjuvant therapy was needed or not has been determined.

High-throughput sequencing, also known as "Next generation" sequencing (NGS), is characterized by sequencing of hundreds of thousands to millions of DNA molecules in parallel, and generally shorter reads.For multiple tumor lesions resected by sMPLC, only biopsy gene information from a single cancer focus may not be enough to identify all active driver gene mutations from the tumor. Therefore, NGS sequencing was proposed for all cancer lesions of sMPLC patients to reflect the full picture of gene mutation in such patients.

The investigators initiated this prospective clinical study to detect lung cancer related genes in tumor tissues and patients with at least 2 tumors that were confirmed as invasive adenocarcinoma by pathology after sMPLC resection (residual non-resectable or non-qualitative pulmonary nodules). At the same time, application of NGS technology to test lung cancer related genes in patients' tumor tissues and blood, patients with lung cancer drive genes were followed up to explore whether different drive genes had an impact on patients' disease progression. In order to investigate the type of gene that causes disease recurrence in patients, tissue or blood test was performed again when disease recurrence occur.

ELIGIBILITY:
Inclusion criteria：

1. Male or female patients: 18-75 years old;
2. ECOG score: 0-1;
3. At least two tumors in patients with invasive lung adenocarcinoma at stage I are pathologically confirmed after sMPLC surgery;
4. Genetic test is performed on the pathological tissues of the tumor lesions excised, and at least one with driver gene;
5. Predicted survival ≥1 year；
6. No more than 3 months after sMPLC surgery (last operation);
7. Good compliance, family members agree to cooperate to receive survival follow-up;
8. Understand and voluntarily sign the informed consent.

Exclusion criteria：

1. Previous or co-existing malignant tumors (patients with resected basal cell carcinoma or other carcinoma in situ are not included);
2. Systemic anti-tumor therapy, including chemotherapy, radiotherapy or targeted therapy (including but not limited to monoclonal antibodies, small-molecule tyrosine kinase inhibitors, etc.) was used before enrollment.
3. Participated in clinical trials of other drugs within 4 weeks
4. All the mutations are insignificant to lung cancer;
5. The investigator is not sure that the subject will be able to complete the study ( management reasons or others).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators initiated this prospective clinical study to detect lung cancer related genes in tumor tissues and patients with at least 2 tumors that were confirmed as invasive adenocarcinoma by pathology after sMPLC resection (residual non-resectable or non-qualitative pulmonary nodules). At the same time, application of NGS technology to test lung cancer related genes in patients' tumor tissues and blood, patients with lung cancer drive genes were followed up to explore whether different drive genes had an impact on patients' disease progression. In order to investigate the type of gene that causes disease recurrence in patients, tissue or blood test was performed again when disease recurrence occur.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-04-22 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
DFS | Two years
  Disease-free survival

SECONDARY OUTCOMES:
Drive-gene about recurrence | Five years
  Explore which drive genes are associated with disease recurrence in patients with different drive genes.

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Jilin University, Changchun, Jilin, China